CLINICAL TRIAL: NCT03791723
Title: Efficacy and Safety of ARNI in Reversing Cardiac Remodeling After Catheter Ablation for Patient With Persistent Atrial Fibrillation and Enlarged Left Atrial
Brief Title: Effect of ARNI in Patients With Persistent AF and Enlarged Left Atrium After Catheter Ablation
Acronym: APART-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, professor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APART-AF
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; Cardiac Remodeling, Atrial; Sacubitril/Valsartan
Keywords: Atrial Fibrillation; Cardiac Remodeling; Sacubitril/Valsartan
MeSH Terms: conditions — Atrial Fibrillation; Atrial Remodeling | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: two groups,group one is for Sacubitril/valsartan 200mg bid or tolerable maximum dose, group two is for valsartan 80mg qd or tolerable maximum dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/valsartan (Experimental): After catheter ablation, during a single blind, run-in period, participants received placebo. Then started with 50 mg sacubitril/valsarta for 2-4 weeks, then uptitrated to 100 mg bid for 2-4 weeks, and thereafter, uptitrated to 200 mg bid or tolerable maximum dose ≥6 months.
  Interventions: Drug: Sacubitril-Valsartan
- Valsartan (Active Comparator): After catheter ablation,during a single blind, run-in period, participants received placebo. Then started with 40mg Valsartan twice daily qd for 2-4 weeks, then were uptitrated to 80mg qd or tolerable maximum dose ≥6 months.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — After catheter ablation,during a single blind, run-in period, participants received placebo. Then started with 50 mg LCZ696 for 2-4 weeks, then uptitrated to 100 mg bid for 2-4 weeks, and thereafter, uptitrated to 200 mg bid or tolerable maximum dose ≥6 months.
  Arms: Sacubitril/valsartan
Drug: Valsartan — After catheter ablation,during a single blind, run-in period, participants received placebo. Then started with 40 mg Valsartan daily (qd) for 2-4 weeks, then were uptitrated to 80mg qd or tolerable maximum dose ≥6 months.
  Arms: Valsartan

SUMMARY:
The purpose of this clinical randomized trial is to evaluate the efficacy and safety of Sacubitril/Valsartan compared with ARB in improving cardiac remodeling in patients With Enlarged Left Atrium Diameter and Persistent AF.

DETAILED DESCRIPTION:
Atrial fibrillation is one of the most common arrhythmia around the word. Prolonged atrial fibrillation may lead to structural changes in the heart such as atrial enlargement, which is an important risk factor for heart failure. Sacubitril/Valsartan is a new drug for the treatment of heart failure, previous studies have shown that it has a good effect in improving cardiac function. For patients with persistent atrial fibrillation and enlarged left atrial, the effect of reversing cardiac remodeling after catheter ablation is unclear. Some studies have described its positive effects in improving cardiac remodeling, but there is still no large-scale randomized controlled trial to further confirm. The investigators hypothesized that Sacubitril/Valsartan can reverse cardiac remodeling in patients with persistent atrial fibrillation and enlarged left atrium compared with ARB after catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent atrial fibrillation undergoing catheter ablation within 2 weeks.
2. ≥18 and ≤75 years of age.
3. Left atrium diameter（LAD）≥35mm, With or without right atrium diameter（RAD）≥40mm，diagnosed by Echocardiographic.
4. patient who are mentally and linguistically able to understand the aim of the trial and to show sufficient compliance in following the trial protocol.
5. Patients receiving ACE inhibitors (ACEI), angiotensin receptor blockers (ARB) and/or a beta blockers must be on a stable dose of these medications stable for the 1 month period prior to Visit.
6. Patients with a controlled systolic BP, defined as a target systolic BP less than 140 mm Hg; participants with BP up to and including 160 mmHg are eligible for enrollment if they are on three or more medications to control BP at randomization.
7. Patients must have an eGFR ≥ 30 ml/min/1.73 m2 at Visit 1 (calculated by the Modification of Diet in Renal Disease formula).
8. Patients with a potassium ≤5.2 mmol/l at Visit 1.

Exclusion Criteria:

1. Patients with prosthetic valves.
2. Any previous LA suigery.
3. Acute coronary syndrome (including MI), cardiac surgery, other major CV surgery within 3 months , or urgent percutaneous coronary intervention within 3 months or and elective PCI within 30 days prior to entry.
4. Presence of hemodynamically significant mitral and /or aortic valve disease.
5. Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic stenosis.
6. Current acute decompensated HF requiring therapy.
7. Allergic to drugs or active ingredients (shakuba, valsartan) or any excipients。
8. Patients with previous history of angioedema associated with ACEI or ARB treatment.
9. Patient with hereditary or idiopathic angioedema.
10. patient with severe liver damage, biliary cirrhosis and cholestasis.
11. Patient with Renal artery stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Left atrial size changes compared to baseline levels | 6months and 12 months
  Echocardiography was used to assess the size of the left atrium, and the changes in atrial structure and baseline levels were compared. The effective index was a gradual decrease in the atrium.

SECONDARY OUTCOMES:
Freedom from AF or AT without the use of antiarrhythmic drugs at 12 months after a single ablation procedure. | 12 months
  Confirmation of atrial fibrillation by electrocardiogram or dynamic electrocardiogram during follow-up. Patients with AF or AT that occurred in the first 3 months after the ablation (blanking period) were censored. Each episode that lasted >30 s was regarded as a recurrence.
all-cause death | 12 months
  all-cause death
Time to first documented recurrence of atrial arrhythmias | 12 months
  Time to first documented recurrence of atrial arrhythmias
Number of hospitalizations caused by heart failure | 12 months
  Number of hospitalizations caused by heart failure
All-cause hospitalizations | 12 months
  All-cause hospitalizations
Number of patients requires adjustment of the drug because of Hypotension | 12 months
  Number of patients requires adjustment of the drug because of Hypotension
Change From Baseline in Echocardiography Parameters: Left Ventricular Ejection Fraction | 12 months
  A limited two-dimensional and Doppler ECHO examination was done to assess ECHO parameters.
Right atrial size changes compared to baseline levels | 12 months
  Echocardiography was used to assess the size of the right atrium, and the changes in atrial structure and baseline levels were compared. The effective index was a gradual decrease in the atrium.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almufleh A, Marbach J, Chih S, Stadnick E, Davies R, Liu P, Mielniczuk L. Ejection fraction improvement and reverse remodeling achieved with Sacubitril/Valsartan in heart failure with reduced ejection fraction patients. Am J Cardiovasc Dis. 2017 Dec 20;7(6):108-113. eCollection 2017. PMID 29348971
- [Result] Januzzi JL, Butler J, Fombu E, Maisel A, McCague K, Pina IL, Prescott MF, Riebman JB, Solomon S. Rationale and methods of the Prospective Study of Biomarkers, Symptom Improvement, and Ventricular Remodeling During Sacubitril/Valsartan Therapy for Heart Failure (PROVE-HF). Am Heart J. 2018 May;199:130-136. doi: 10.1016/j.ahj.2017.12.021. Epub 2018 Feb 13. PMID 29754651